CLINICAL TRIAL: NCT06745128
Title: Tirzepatide for Individuals With Comorbid Obesity and Methamphetamine Use Disorder
Brief Title: Tirzepatide for Obesity and Meth Use Disorder
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Manish Jha, MBBS, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2024-1221
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Obesity; Methamphetamine Use Disorder
Keywords: Methamphetamine; Methamphetamine Use Disorder; MUD; Overweight; Obesity; Tirzepatide; Weight management
MeSH Terms: conditions — Obesity; Overweight | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tirzepatide (Experimental): Eligible participants who are enrolled will receive once-weekly subcutaneous injections of tirzepatide for a 32-week period in accordance with FDA-prescribing label guidelines.
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Eligible participants who are enrolled will receive once-weekly subcutaneous injections of tirzepatide for a 32-week period. Following the instructions of the FDA-approved prescribing label, participants or a licensed study clinician will administer the tirzepatide injection subcutaneously in either the abdomen, thigh, or upper arm once weekly for 32 weeks total. Following the instructions of the FDA-approved prescribing label, the dosing schedule will include a 4-week titration at a starting dosage of 2.5mg/week. After four weeks, dosage will be increased in 2.5mg increments. The recommended maintenance dosages per prescribing label are 5mg/week, 10mg/week, or 15mg/week injected subcutaneously. Maximum dosage (up to 15mg/week) will be optimized for each individual. We will use commercially available tirzepatide, primarily dispensed as ZEPBOUND® for this study, but in the event of medication shortage or other pharmacy-related issue, MOUNJARO® may be dispensed as an alternative.
  Other Names: ZEPBOUND; MOUNJARO

SUMMARY:
This is an open-label pilot study to evaluate the feasibility and preliminary efficacy of using tirzepatide when prescribed for its United States (US) Food and Drug Administration (FDA)-approved weight-related indication in individuals with comorbid methamphetamine use disorder.

DETAILED DESCRIPTION:
This study will enroll up to 45 individuals with moderate-to-severe methamphetamine use disorder who meet the FDA-approved weight-related indication for tirzepatide [as an adjunct to a reduced-calorie diet and increased physical activity for chronic weight management in adults with an initial body mass index (BMI) of: 1) 30 kg/m2 or greater (obesity) or 2) 27 kg/m2 or greater (overweight) in the presence of at least one weight-related comorbid condition (e.g., hypertension, dyslipidemia, type 2 diabetes mellitus, obstructive sleep apnea or cardiovascular disease)].

Enrolled participants will receive weekly treatment with tirzepatide for a 32-week period that will be followed by 4-week-long observational follow-up. Participants of this study will be seen for weekly visits where they will complete clinical and/or laboratory assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 to 65 years of age, inclusive.
2. Be able to provide informed consent and ask relevant questions.
3. Stated willingness to comply with all study procedures and availability for the duration of the study.
4. Be willing to adhere to the study medication regimen
5. Meet DSM-5 criteria for moderate or severe methamphetamine use disorder.
6. Self-report methamphetamine use on 18 or more days in the 30-day period prior to written informed consent using the Timeline Followback (TLFB).
7. Have an initial body mass index (BMI) at screening of:

   1. 30 kg/m2 or greater (obesity)
   2. 27 kg/m2 or greater (overweight) in the presence of at least one weight-related comorbid condition (e.g., hypertension, dyslipidemia, type 2 diabetes mellitus, obstructive sleep apnea or cardiovascular disease).
8. If biologically female and is or becomes sexually active with a biological male, must agree to use acceptable methods of contraception and have urine pregnancy testing during participation in the study, unless unable to get pregnant

   a. Appropriate birth control methods include: i. Oral contraceptives, contraceptive patch, hormonal vaginal contraceptive ring (with restrictions related to dose change given the medication interactions between tirzepatide and oral contraceptives).

   ii. Barrier (diaphragm or condom) iii. Contraceptive implant iv. Medroxyprogesterone acetate injection v. Intra-uterine device vi. Complete abstinence from sexual intercourse vii. Surgical sterilization
9. Agreement to adhere to Lifestyle Considerations (see section 5.3) throughout study duration

Exclusion Criteria:

1. Current or recent use (within 3 months prior to consent) of other tirzepatide-containing products or any other GLP-1 receptor agonist
2. Current or recent use (within 30 days) of sulfonylureas, other concomitantly administered insulin secretagogue, or insulin
3. Current or recent use (within 3 months prior to consent) of other weight loss agents
4. Weight loss surgery within 12 months prior to consent
5. Current eating disorder per clinician evaluation
6. Personal or family history of Medullary Thyroid Carcinoma
7. History of Multiple Endocrine Neoplasia syndrome type 2
8. Known serious hypersensitivity (e.g., anaphylaxis, angioedema) to tirzepatide or any of the excipients in tirzepatide
9. History of angioedema or anaphylaxis with a GLP-1 receptor agonist
10. Current Stage 3 or higher Chronic Kidney Disease, defined as eGFR <60 at Screening
11. Current inadequately controlled diabetes, defined as HbA1c > 7.0 at Screening
12. History of diabetic retinopathy
13. Current pregnancy or lactation
14. Treatment with another investigational drug or intervention within the past one month (30 days prior to consent)
15. Have any condition for which study participation would not be in their best interest (e.g., cognitive impairment, unstable general medical condition, intoxication, active psychosis) or that could prevent, limit, or confound the protocol-specified assessments, in the opinion of the investigator or their designee.
16. Require immediate hospitalization for psychiatric disorder or suicidal risk as assessed by a licensed study clinician.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Effect of tirzepatide on self-reported use of methamphetamine | 36 weeks
  Self-reported use of methamphetamine will be assessed through Timeline Followback. The Timeline Followback procedure will be used to elicit the participant's self-reported use of illicit substances, including but not limited to stimulants, and polysubstance use starting at the Screening Visit and continuing throughout study participation. During the Screening Visit, this form will be used to assess illicit use of substances for the 30-day period prior to written consent. During the study, TLFB will be administered to document the participant's self-reported use of illicit substances, nicotine, and tobacco for each visit since the previous TLFB assessment. Participant's drug of choice will be asked and determined by study coordinator and recorded along with the TLFB assessment.

SECONDARY OUTCOMES:
Feasibility of using tirzepatide in individuals with Methamphetamine Use Disorder | 4 weeks
  Feasibility will be defined as the number of participants who receive a dose of tirzepatide of at least a 5mg/week for at least four weeks.
Changes in body mass index from baseline to the end of the 32-week treatment phase | 32 weeks
  Body mass index will be calculated using measurements of height and weight.
Changes in self-reported symptoms of anhedonia from baseline to the end of the 32-week treatment phase | 32 weeks
  Anhedonia, the inability to experience pleasure, will be assessed by the Snaith-Hamilton Pleasure Scale (SHAPS). The SHAPS questionnaire contains 14 items related to experiencing pleasure over the last several days. Participants are asked to rate their level of agreement or disagreement with each prompt. The scale has a scoring range of 0-14 where a higher point value indicates a higher level of anhedonia.
Changes in High-sensitivity C-reative protein (hs-CRP) levels from baseline to the end of the 32-week treatment phase | 32 weeks
  Clinical laboratory assessments for High-Sensitivity C-Reactive Protein (HsCRP) test will be performed to help determine eligibility at screening and monitor participant's overall health condition.
Changes in gastrointestinal symptom severity from baseline until the end of the 32-week treatment phase | 32 weeks
  Gastrointestinal symptom severity will be assessed by the Gastrointestinal Symptom Rating Scale (GSRS): a disease-specific instrument of 15 items combined into five symptom clusters depicting Reflux, Abdominal pain, Indigestion, Diarrhea and Constipation. The GSRS scale is graded on a seven-point Likert-type scale where a lower score (1) represents less symptom severity and highest score (7) represents greater symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Manish Jha, M.B.B.S., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data is planned to be shared with other researchers.

REFERENCES:
- [Background] Volkow ND, Xu R. GLP-1R agonist medications for addiction treatment. Addiction. 2025 Feb;120(2):198-200. doi: 10.1111/add.16626. Epub 2024 Jul 24. PMID 39049203
- [Background] Lahteenvuo M, Tiihonen J, Solismaa A, Tanskanen A, Mittendorfer-Rutz E, Taipale H. Repurposing Semaglutide and Liraglutide for Alcohol Use Disorder. JAMA Psychiatry. 2025 Jan 1;82(1):94-98. doi: 10.1001/jamapsychiatry.2024.3599. PMID 39535805
- [Background] Coffin PO, Suen LW. Methamphetamine Toxicities and Clinical Management. NEJM Evid. 2023 Dec;2(12):EVIDra2300160. doi: 10.1056/EVIDra2300160. Epub 2023 Nov 28. PMID 38320504
- [Background] Kulich KR, Madisch A, Pacini F, Pique JM, Regula J, Van Rensburg CJ, Ujszaszy L, Carlsson J, Halling K, Wiklund IK. Reliability and validity of the Gastrointestinal Symptom Rating Scale (GSRS) and Quality of Life in Reflux and Dyspepsia (QOLRAD) questionnaire in dyspepsia: a six-country study. Health Qual Life Outcomes. 2008 Jan 31;6:12. doi: 10.1186/1477-7525-6-12. PMID 18237386
- [Background] Tan B, Pan XH, Chew HSJ, Goh RSJ, Lin C, Anand VV, Lee ECZ, Chan KE, Kong G, Ong CEY, Chung HC, Young DY, Chan MY, Khoo CM, Mehta A, Muthiah MD, Noureddin M, Ng CH, Chew NWS, Chin YH. Efficacy and safety of tirzepatide for treatment of overweight or obesity. A systematic review and meta-analysis. Int J Obes (Lond). 2023 Aug;47(8):677-685. doi: 10.1038/s41366-023-01321-5. Epub 2023 May 31. PMID 37253796
- [Background] Barry D, Clarke M, Petry NM. Obesity and its relationship to addictions: is overeating a form of addictive behavior? Am J Addict. 2009 Nov-Dec;18(6):439-51. doi: 10.3109/10550490903205579. PMID 19874165
- [Background] Franken IH, Rassin E, Muris P. The assessment of anhedonia in clinical and non-clinical populations: further validation of the Snaith-Hamilton Pleasure Scale (SHAPS). J Affect Disord. 2007 Apr;99(1-3):83-9. doi: 10.1016/j.jad.2006.08.020. Epub 2006 Sep 20. PMID 16996138
- [Background] Sobell LC, Sobell MB, Leo GI, Cancilla A. Reliability of a timeline method: assessing normal drinkers' reports of recent drinking and a comparative evaluation across several populations. Br J Addict. 1988 Apr;83(4):393-402. doi: 10.1111/j.1360-0443.1988.tb00485.x. No abstract available. PMID 3395719